CLINICAL TRIAL: NCT07214467
Title: Individualized Adaptive Deep Brain Stimulation in Opioid Use Disorder
Acronym: aDBS OUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Khaled Moussawi, MD, PhD, Associate Professor in Residence, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-43357
Record Dates: First submitted 2025-09-25; First posted 2025-10-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorder (SUD); Opioid Use Disorder (OUD)
Keywords: Opioid; SUD; OUD; Substance Use; Substance Use Disorder; Addiction; Opioid Use Disorder; Opioid Use; deep brain stimulation; Neuromodulation; stereo-EEG; brain mapping
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Behavior, Addictive | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, sham controlled Latin square design, followed by open label follow up period pilot trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All study participants and study personnel involved in clinical outcomes collection and analysis will be blinded. Study personnel overseeing participant safety, randomization, and DBS optimization will not be blinded and will not be involved in assessing the clinical outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- aDBS / cDBS / sham Stimulation (Other): Participants in this group will first receive adaptive deep brain stimulation (aDBS), followed by continuous deep brain stimulation (cDBS), and finally a sham stimulation. Each period of the randomized controlled trial (aDBS, cDBS, and sham) will last 4 months.
  Interventions: Device: Deep Brain Stimulation
- sham / aDBS / cDBS (Other): Participants in this group will first receive sham stimulation, followed by adaptive deep brain stimulation (aDBS), and finally continuous deep brain stimulation (cDBS). Each period of the randomized controlled trial (aDBS, cDBS, and sham) will last 4 months.
  Interventions: Device: Deep Brain Stimulation
- cDBS / sham / aDBS (Other): Participants in this group will first receive continuous deep brain stimulation (cDBS), followed by sham stimulation, and finally adaptive deep brain stimulation (aDBS). Each period of the randomized controlled trial (aDBS, cDBS, and sham) will last 4 months.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — An individualized aDBS protocol will be used to examine therapeutic effect.
  Other Names: DBS

SUMMARY:
The purpose of this study is to determine if personalized (adaptive) Deep Brain Stimulation (DBS) based upon invasive brain mapping is safe and can lead to better outcomes like reductions in craving and opioid use.

DETAILED DESCRIPTION:
This study will enroll individuals with severe Opioid Use Disorder (OUD) who have not responded to standard treatments. The devices used in this study are investigational, which means they are not approved by the Food and Drug Administration (FDA) to treat OUD. The information we obtain in this study will be used to better understand the mechanisms of OUD in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Adults (all genders) 22 to 75 years old.
* Current diagnosis of severe primary opioid use disorder (OUD) (>= 6 on DSM-5 OUD criteria) (any form of opioid use).
* History of opioid use for more than 5 years.
* Participants are seeking treatment for their OUD.
* Participants have insight into their opioid use disorder (score > 26 on the recognition subscale of the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES V.8))
* OUD is treatment refractory: unable to achieve sustained remission over the past 5 years, despite at least three treatment attempts (outpatient, residential, inpatient), with at least one treatment attempt involving taking a first-line medication for OUD (MOUD) such as buprenorphine, methadone, or extended-release naltrexone. Treatment failure is defined as continued opioid use or relapse during or after completion of treatment. Sustained remission is defined per DSM-5 as not meeting any OUD criteria except craving for > 12 months. Documented adherence: participants must have documented adherence to the failed first-line MOUD for at least 8 weeks (PMID: 29083570).
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Social support system and stable living arrangement to provide assurances that the subject will adhere to study requirements: family or friends who live with or near the subject, and can provide collateral information, monitor the subject's behavior, support, and encourage the subject to participate in follow-up visits and evaluations.
* For individuals of reproductive potential: use of highly effective contraception for at least 4 weeks prior to sEEG surgery and agreement to use such a method during study participation.

Exclusion Criteria:

* Pregnancy or lactation.
* Non-English speaking.
* Participants are not willing to start MOUD treatment with buprenorphine or to switch MOUD to buprenorphine if they are already on other MOUD, for the duration of the study.
* OUD treatment with another investigational drug or other intervention within 3 months.
* History of primary psychosis or Bipolar I disorder per the medical interview.
* History of severe personality disorder that could interfere with study participation (e.g., antisocial personality disorder) per the medical interview.
* History of traumatic brain injury with loss of consciousness greater than 5 minutes.
* Clinically significant cognitive impairment per neuropsychological testing.
* History of suicidal attempts in the past 3 years or current suicidal thoughts per psychiatric evaluation.
* Coagulopathy: INR > 1.4, aPTT > 40 s, platelets < 100,000.
* Current clinically significant medical or neurologic disease that affects brain function (e.g., recent stroke, myocardial infarction, seizures not due to alcohol withdrawal).
* Clinically significant abnormality on structural brain MRI scan.
* Life expectancy less than 24 months per the clinical judgment of study investigators (e.g., terminal cancers).
* Any labeled DBS contraindication or inability to have brain MRI: certain pacemakers, metal in body, inability to undergo awake operation, significant cardiac or other medical risk factors for surgery, infection, and coagulopathy.
* Exclusion for early remission: participants who achieve early remission after initiating buprenorphine during the screening phase (prior to the sEEG phase) will be excluded from the study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2031-11-22 (Estimated); Study Completion 2031-11-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events during sEEG phase | Up to 2 weeks during sEEG phase.
  To assess the safety of sEEG mapping in patients with severe and refractory OUD.
Incidence of adverse events during aDBS phase | Up to 16 months from time of DBS implantation.
  To assess the safety of aDBS in patients with severe and refractory OUD.

SECONDARY OUTCOMES:
sEEG Mapping: Brain mapping | Up to 2 weeks during sEEG phase.
  To identify individualized brain targets for sensing neural biomarkers of craving and stimulation to mitigate craving.
Opioid use duirng aDBS treatment | Up to 16 months from time of DBS implantation.
  To evaluate the preliminary efficacy of individualized aDBS in patients with severe and refractory OUD by measuring the effects of aDBS on opioid use measured with TLFB.
Overall functioning duirng aDBS treatment | Up to 16 months from time of DBS implantation.
  To evaluate the preliminary efficacy of individualized aDBS in patients with severe and refractory OUD by measuring the effects of aDBS on quality of life measured with SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Moussawi, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou H, Xu J, Jiang J. Deep brain stimulation of nucleus accumbens on heroin-seeking behaviors: a case report. Biol Psychiatry. 2011 Jun 1;69(11):e41-2. doi: 10.1016/j.biopsych.2011.02.012. Epub 2011 Apr 13. No abstract available. PMID 21489407
- [Background] Chen L, Li N, Ge S, Lozano AM, Lee DJ, Yang C, Li L, Bai Q, Lu H, Wang J, Wang X, Li J, Jing J, Su M, Wei L, Wang X, Gao G. Long-term results after deep brain stimulation of nucleus accumbens and the anterior limb of the internal capsule for preventing heroin relapse: An open-label pilot study. Brain Stimul. 2019 Jan-Feb;12(1):175-183. doi: 10.1016/j.brs.2018.09.006. Epub 2018 Sep 14. PMID 30245163
- [Background] Rezai AR, Mahoney JJ, Ranjan M, Haut MW, Zheng W, Lander LR, Berry JH, Farmer DL, Marton JL, Tirumalai P, Mears A, Thompson-Lake DGY, Finomore VS, D'Haese PF, Aklin WM, George DT, Corrigan JD, Hodder SL. Safety and feasibility clinical trial of nucleus accumbens deep brain stimulation for treatment-refractory opioid use disorder. J Neurosurg. 2023 Jun 9;140(1):231-239. doi: 10.3171/2023.4.JNS23114. Print 2024 Jan 1. PMID 37329519
- [Background] Kuhn J, Moller M, Treppmann JF, Bartsch C, Lenartz D, Gruendler TO, Maarouf M, Brosig A, Barnikol UB, Klosterkotter J, Sturm V. Deep brain stimulation of the nucleus accumbens and its usefulness in severe opioid addiction. Mol Psychiatry. 2014 Feb;19(2):145-6. doi: 10.1038/mp.2012.196. Epub 2013 Jan 22. No abstract available. PMID 23337942